CLINICAL TRIAL: NCT00182442
Title: A One-Year Multi-Centre Randomized, Double Blind, Controlled Effectiveness Study of Quetiapine and Olanzapine, Comparing Their Relative Potential in Improving Neuro-Cognitive Deficits, Functional Outcomes and Quality of Life in Schizophrenia
Brief Title: Cognition, Functioning and Quality of Life
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: AstraZeneca (Industry)
Organization: McMaster University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 02-2179
Record Dates: First submitted 2005-09-14; First posted 2005-09-16 (Estimated); Last update posted 2006-10-11 (Estimated); Status verified 2005-03

CONDITIONS: Schizophrenia
Keywords: Cognitive deficits; Psychosocial functioning; Quality of Life
MeSH Terms: conditions — Schizophrenia; Cognition Disorders | interventions — Olanzapine; Quetiapine Fumarate

INTERVENTIONS:
Drug: Olanzapine & Quetiapine

SUMMARY:
People affected by schizophrenia often experience poor concentration, lapses in memory and difficulty with completing tasks; and this set of problems are known as neuro-cognitive deficits. Traditional medications used in the treatment of schizophrenia have not been particularly useful in improving these problems, while the recently introduced medications are expected to be superior in this respect. The proposed research study is designed to assess the effect of two of the new medications (Zyprexa and Seroquel) in improving the neurocognitive deficits associated with schizophrenia.

DETAILED DESCRIPTION:
Schizophrenia is a chronic, debilitating psychiatric disorder with complex clinical presentation, partially responsiveness to treatment and varied outcomes. Though modern anti-psychotic drugs have been used to treat the illness for the past 50 years, it has been consistently observed that a significant proportion of people diagnosed with schizophrenia do not respond adequately to these medications. Even among those people who show symptomatic improvement, the benefit does not translate into improved functioning in real life setting.

Research in the past 10 years revealed two significant findings: 1) it is now known that a proportion of people with schizophrenia have neurocognitive deficits as part of their clinical profile. Neuro-cognitive deficits refer to impairments in attention, concentration, memory, use of language, decision making and subtle aspects of judgment. 2) Traditional antipsychotic drugs have not been useful in improving neurocognitive deficits, while claims have been made that novel antipsychotic drugs (Quetiapine, Olanzapine and Risperidone) may have some beneficial effects in improving the neurocognitive deficits associated with schizophrenia. In an earlier investigation, we have noticed that Quetiapine produced clinically significant improvement in neurocognitive deficits compared to other antipsychotic drugs; and there have been two additional reports confirming this distinctive advantage of Quetiapine.

Based on these preliminary results, the present study is designed to address the following questions. 1) To examine whether the neurocognitive deficits associated with schizophrenia have an impact on the community functioning and quality of life of individuals affected by this illness, and 2) whether Quetiapine (Seroquel) is significantly more effective than Olanzapine (Zyprexa) in improving neurocognitive deficits, community functioning and quality of life.

The study sample will include a total of 120 patients with the diagnosis of schizophrenia or schizoaffective disorder, who will require antipsychotic drug treatment. The sample size calculation is based on the expected differences between the two compared medications, in terms of their ability to improve the neurocognitive cluster score on PANSS (Positive and negative symptoms scale) detected in our earlier study.The study is designed as a prospective double-blind, randomized controlled trial, using Quetiapine and Olanzapine as drugs for comparison. Eligible participants will undergo a baseline clinical and neurocognitive evaluation and randomly assigned to receive either Quetiapine or Olanzapine treatment. Both patients and controls are blinded to the nature of the medication being prescribed. However, the clinicians will have the flexibility to increase the dose as clinically appropriate. The goal is to achieve symptom stability and monitor the progress in community functioning, and changes in perceived quality of life. The participants will continue with the medication at least for a period of one year, and the outcome evaluations will be performed at 1, 3, 6, 9 and 12 month points. These include re-assessment of clinical symptoms and neurocognitive deficits and community functioning, using appropriate measurement tools.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia confirmed by administering SCID and,
* Subjects consecutively referred for optimizing antipsychotic drug therapy, i.e. a change of medication from conventional medications or Risperidone is indicated due to lack of efficacy, side-effects or poor subjective tolerability.
* Competent to provide an informed consent.

Exclusion Criteria:

* Substance dependence, mental retardation, head injury or other primary neurological disorders.
* Imminent risk due to suicidal or aggressive behavior (a score of five or more on the hostility item on the PANSS).
* A pattern of social instability, which could hamper long-term follow-up.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80
Dates: Start 2003-10; Study Completion 2006-03

PRIMARY OUTCOMES:
Primary outcome measures include changes in neurocognitive test scores, changes in measures of community functioning and quality of life.

SECONDARY OUTCOMES:
Secondary outcomes include changes in treatment adherence, subjective satisfaction with antipsychotic drug therapy, clinical symptoms and side effects.

CONTACTS AND LOCATIONS:
Overall Officials: Lakshmi P Voruganti, MD, Principal Investigator — McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada